CLINICAL TRIAL: NCT03440554
Title: Non-contrast MR Imaging for Whole Body Cancer Detection and Characterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Prostate Cancer Foundation (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Hahn, Assistant Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 151686
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Restriction spectrum imaging; Magnetic resonance imaging; MRI; RSI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prostate cancer patients will have a research whole body MRI scan within 90 days of their standard of care imaging. Patients receiving additional standard of care imaging within 12 months of the research scan will be asked to have an additional research scan within 90 days of their follow-up imaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Whole Body Non-Contrast MRI (Experimental)
  Interventions: Diagnostic Test: Whole Body Non-Contrast MRI

INTERVENTIONS:
Diagnostic Test: Whole Body Non-Contrast MRI — Whole Body Non-Contrast MRI in Prostate Cancer Patients

SUMMARY:
This study aims to learn how to improve MRIs (Magnetic Resonance Imaging) that do not require the patient to be injected with a contrast dye. Researchers expect to learn how to better find and describe tumors in patients with prostate cancer. Participants have a whole body research MRI scan within 90 days of a standard-of-care imaging procedure. The research study will collect copies of those scans to compare to the research scans as part of the study analysis.

Patients who have additional standard-of-care scans within 12 months after their research scan may be asked to have a second non-contrast MRI for research within 90 days of their follow-up standard of care imaging. The whole body MRI scan will be compared to the standard-of-care scan for prostate cancer detection and to assess patient response to standard-of-care treatment.

DETAILED DESCRIPTION:
Participants will undergo a whole body non-contrast MRI study with a whole-body protocol incorporating routine clinical sequences as well as non-contrast research sequences. The patient will also undergo clinically indicated standard-of-care imaging such as PET/CT, CT, Technetium-99m bone scan or MRI with contrast as determined by the patient's oncologist. When the standard-of-care imaging has not yet been performed upon enrollment, the research MRI will ideally be performed on the same day as the standard-of-care exam. However, scheduling constraints and patient time constraints may preclude scheduling both scans on the same day. In this case, the scans will be performed within a week 90 days of each other. An experienced radiologist will read both scans and results will be provided to the patient's oncologist for clinical follow up.

Patients receiving additional standard-of-care imaging within 12 months after the research MRI may be asked to return for an additional whole body MRI scan within 90 days of their standard-of-care scan. The additional research scan will be requested of patients that have evidence of progression during ongoing standard of care treatment and monitoring. The additional scan would be requested of those patients to compare baseline scans to those that are completed during standard of care imaging. This would be an additional tool to verify disease progression or treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have known or suspected genitourinary metastatic disease and have already had or will have a CT, PET/CT, bone scan or MRI with contrast.
* Age ≥ 18 years.
* ECOG performance status 0-3.
* Capacity to give informed consent.
* Ability to lay supine for 30-60 minutes
* Ability to hear adequately without hearing aids.

Exclusion Criteria:

* Patients with medical implants/devices or indwelling foreign material considered unsafe for MRI scanning will be excluded. Safety of medical implants/devices will be determined by the current UC San Diego Radiology and Imaging Services MRI safety policy. The name, manufacturer, and model number of any medical implant/device contained within a potential study subject will be obtained and reviewed to determine safety. Patients will be excluded if any implant/device is found to be unsafe for MRI scanning.
* Patients may be excluded if their weight exceeds 350 lbs, the limit for the safe operation of the MRI scanning table.
* A patient who is pregnant or trying to become pregnant will be excluded.
* Patients with any other condition that, in the opinion of the investigator, may deem them ineligible for study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Specificity and Sensitivity of Whole Body MRI in Relation to Standard-of-Care Imaging | 15 months
  Paired t-test
Covariance of Whole Body MRI Cellularity Index (CI) and PET/CT Standardized Uptake Value (SUV) | 15 months
  For each identified lesion in the PET/CT, the lesion will be outlined, the size measured in millimeters, and the SUV will be calculated using the following equation:
  SUV= (decay-(corrected activity (kBq))/(tissue volume (ml) ))/(injected=(FDG activity (kBq))/(body weight (g) ))
  Baseline SUVs will also be calculated within normal appearing tissue.
  Similarly, for each identified lesion in the whole-body RSI-MRI, the lesion will be outlined, the size measured as indicated above, and the CI will be calculated. Baseline CIs will also be calculated within normal appearing tissue.
  The quantitative data will be analyzed for correlation across all lesions in all patients to determine the degree to which PET/CT SUV values and RSI-MRI CI values co-vary. Significance of the correlation coefficient, compared to zero correlation, will be assessed via the Student t-test, with alpha set to 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Hahn, MD, Principal Investigator — UC San Diego Moores Cancer Center
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marusyk A, Almendro V, Polyak K. Intra-tumour heterogeneity: a looking glass for cancer? Nat Rev Cancer. 2012 Apr 19;12(5):323-34. doi: 10.1038/nrc3261. PMID 22513401
- [Background] Jacobs EL, Haskell CM. Clinical use of tumor markers in oncology. Curr Probl Cancer. 1991 Nov-Dec;15(6):299-360. doi: 10.1016/0147-0272(91)90005-u. PMID 1760927
- [Background] Drukteinis JS, Mooney BP, Flowers CI, Gatenby RA. Beyond mammography: new frontiers in breast cancer screening. Am J Med. 2013 Jun;126(6):472-9. doi: 10.1016/j.amjmed.2012.11.025. Epub 2013 Apr 3. PMID 23561631
- [Background] Fischer AH. The diagnostic pathology of the nuclear envelope in human cancers. Adv Exp Med Biol. 2014;773:49-75. doi: 10.1007/978-1-4899-8032-8_3. PMID 24563343
- [Background] White NS, McDonald C, Farid N, Kuperman J, Karow D, Schenker-Ahmed NM, Bartsch H, Rakow-Penner R, Holland D, Shabaik A, Bjornerud A, Hope T, Hattangadi-Gluth J, Liss M, Parsons JK, Chen CC, Raman S, Margolis D, Reiter RE, Marks L, Kesari S, Mundt AJ, Kane CJ, Carter BS, Bradley WG, Dale AM. Diffusion-weighted imaging in cancer: physical foundations and applications of restriction spectrum imaging. Cancer Res. 2014 Sep 1;74(17):4638-52. doi: 10.1158/0008-5472.CAN-13-3534. PMID 25183788
- [Background] Attariwala R, Picker W. Whole body MRI: improved lesion detection and characterization with diffusion weighted techniques. J Magn Reson Imaging. 2013 Aug;38(2):253-68. doi: 10.1002/jmri.24285. PMID 23960006
- [Background] White NS, Dale AM. Distinct effects of nuclear volume fraction and cell diameter on high b-value diffusion MRI contrast in tumors. Magn Reson Med. 2014 Nov;72(5):1435-43. doi: 10.1002/mrm.25039. Epub 2013 Dec 19. PMID 24357182
- [Background] White NS, Leergaard TB, D'Arceuil H, Bjaalie JG, Dale AM. Probing tissue microstructure with restriction spectrum imaging: Histological and theoretical validation. Hum Brain Mapp. 2013 Feb;34(2):327-46. doi: 10.1002/hbm.21454. Epub 2012 Jan 16. PMID 23169482
- [Background] Rakow-Penner RA, White NS, Parsons JK, Choi HW, Liss MA, Kuperman JM, Schenker-Ahmed N, Bartsch H, Mattrey RF, Bradley WG, Shabaik A, Huang J, Margolis DJ, Raman SS, Marks L, Kane CJ, Reiter RE, Karow DS, Dale AM. Novel technique for characterizing prostate cancer utilizing MRI restriction spectrum imaging: proof of principle and initial clinical experience with extraprostatic extension. Prostate Cancer Prostatic Dis. 2015 Mar;18(1):81-5. doi: 10.1038/pcan.2014.50. Epub 2015 Jan 6. PMID 25559097
- [Background] White NS, McDonald CR, Farid N, Kuperman JM, Kesari S, Dale AM. Improved conspicuity and delineation of high-grade primary and metastatic brain tumors using "restriction spectrum imaging": quantitative comparison with high B-value DWI and ADC. AJNR Am J Neuroradiol. 2013 May;34(5):958-64, S1. doi: 10.3174/ajnr.A3327. Epub 2012 Nov 8. PMID 23139079
- [Background] Liss MA, White NS, Parsons JK, Schenker-Ahmed NM, Rakow-Penner R, Kuperman JM, Bartsch H, Choi HW, Mattrey RF, Bradley WG, Shabaik A, Huang J, Margolis DJ, Raman SS, Marks LS, Kane CJ, Reiter RE, Dale AM, Karow DS. MRI-Derived Restriction Spectrum Imaging Cellularity Index is Associated with High Grade Prostate Cancer on Radical Prostatectomy Specimens. Front Oncol. 2015 Feb 17;5:30. doi: 10.3389/fonc.2015.00030. eCollection 2015. PMID 25741473
- [Background] McCammack KC, Kane CJ, Parsons JK, White NS, Schenker-Ahmed NM, Kuperman JM, Bartsch H, Desikan RS, Rakow-Penner RA, Adams D, Liss MA, Mattrey RF, Bradley WG, Margolis DJ, Raman SS, Shabaik A, Dale AM, Karow DS. In vivo prostate cancer detection and grading using restriction spectrum imaging-MRI. Prostate Cancer Prostatic Dis. 2016 Jun;19(2):168-73. doi: 10.1038/pcan.2015.61. Epub 2016 Jan 12. PMID 26754261
- [Derived] Conlin CC, Feng CH, Digma LA, Rodriguez-Soto AE, Kuperman JM, Rakow-Penner R, Karow DS, White NS, Seibert TM, Hahn ME, Dale AM. A Multicompartmental Diffusion Model for Improved Assessment of Whole-Body Diffusion-weighted Imaging Data and Evaluation of Prostate Cancer Bone Metastases. Radiol Imaging Cancer. 2023 Jan;5(1):e210115. doi: 10.1148/rycan.210115. PMID 36705559